CLINICAL TRIAL: NCT04462562
Title: The Diagnostic Performance Assessment of Quantitative Ultrasound Imaging Indices for Differentiating Hepatic Steatosis Grade in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Quantitative US for Evaluation of Hepatic Steatosis in NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medison (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH 2002-020-1099
Record Dates: First submitted 2020-03-31; First posted 2020-07-08 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Fatty Liver; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quantitative ultrasound imaging parameters (Experimental): quantitative ultrasound imaging parameters
  * tissue attenuation imaging (TAI) parameter
  * tissue scatter-distribution imaging (TSI) parameter
  * Hepatorenal index (semi-auto, EzHRI)
  Interventions: Diagnostic Test: Quantitative US (Samsung Medison, RS85A)

INTERVENTIONS:
Diagnostic Test: Quantitative US (Samsung Medison, RS85A) — In each patients, measurements of tissue attenuation imagine (TAI), tissue scatter-distribution imaging (TSI) parameters, hepatorenal index (EzHRI) will be performed

SUMMARY:
The purpose of this study is to evaluate diagnostic performance of quantitative ultrasonographic parameters for the assessment of hepatic steatosis with find optimal cut-off values in patients with non-alcoholic fatty liver disease using magnetic resonance imaging proton density fat fraction (MRI-PDFF) and MR spectroscopy as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* patients with known NAFLD or suspected of having NAFLD
* Patients who are scheduled hepatectomy for living donor liver donation
* aged ≥ 18 years who are willing and able to complete all procedures

Exclusion Criteria:

* excessive alcohol consumption within 2 years (40g/day for men, 20g/day for women)
* clinical, laboratory, or histologic evidence of a liver disease other than NAFLD, including viral hepatitis, autoimmune hepatitis, or genetic or acquired disorders
* use of steatogenic or hepatotoxic medication
* evidence of decompensated liver disease
* history of liver surgery
* contraindication to MRI
* any other condition believed by investigator to affect a patients' compliance, or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (area under the ROC curve (AUC)) of quantitative US (QUS) parameters (TAI, TSI) for detection of fatty liver (MRI-PDFF 5 percent) | 1 month
  Reference standard: MRI-proton density fat fraction or MR spectroscopy value (5 percent)
  - ROC curve analysis of each QUS parameters (TAI, TSI, EzHRI) for the detection of MRI-PDFF >5 percent patients

SECONDARY OUTCOMES:
Diagnostic performance (area under the ROC curve (AUC)) of QUS parameters (TAI, TSI) for detection of moderate fatty liver (MRI-PDFF 10, 20 percent) | 1 month
  Reference standard: MRI-PDFF or MR spectroscopy value (10 percent, 15 percent, 15 percent, 20 percent, 25 percent)
  - ROC curve analysis of each QUS parameters (TAI, TSI, EzHRI) for the detection of MRI-PDFF >10, >20 percent patients
Correlation of QUS parameters and MR fat fraction | 1 month
  reference standard: MRI-PDFF or MR spectroscopy value (percent)
  - spearman's rank correlation of QUS parameters (TAI, TSI) values with MR fat fraction(percent)
Intra-observer agreement of quantitative US parameters | 1 day
  Intraclass correlation coefficient (ICC), coefficient of variation (CV) of QUS parameter values (TAI value, TSI value)
Correlation between estimated fat fraction from deep learning model and MRI-proton density fat fraction | 1 month
  pearson correlation coefficient (r) between estimated fat fraction and MRI-proton density fat fraction
Diagnostic performance (area under the ROC curve (AUC)) of deep leraning model using QUS parametric maps for detection fatty liver (10 percent, 15 percent, 15 percent, 20 percent) | 1 month
  Reference standard: MRI-proton density fat fraction (10 percent, 15 percent, 20 percent, 20 percent)
Diagnostic performance (area under the ROC curve (AUC)) of deep leraning model using QUS parametric maps for detection fatty liver (5 percent) | 1 month
  Reference standard: MRI-proton density fat fraction (5 percent)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jeon SK, Lee JM, Joo I, Yoon JH, Lee G. Two-dimensional Convolutional Neural Network Using Quantitative US for Noninvasive Assessment of Hepatic Steatosis in NAFLD. Radiology. 2023 Apr;307(1):e221510. doi: 10.1148/radiol.221510. Epub 2023 Jan 3. PMID 36594835